CLINICAL TRIAL: NCT04946526
Title: Bioavailability of Sulforaphane From a Glucoraphanin-Rich Broccoli Seed Supplement With or Without Added Myrosinase From Mustard Seed Powder
Brief Title: Broccoli Sulforaphane Bioavailability With Mustard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Brassica Foundation for Chemoprotection Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-0216
Record Dates: First submitted 2021-06-17; First posted 2021-07-01 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Sulforaphane Bioavailability
Keywords: broccoli; mustard; sulforaphane; glucoraphanin; bioavailability

STUDY DESIGN:
Intervention Model Description: Randomized crossover with a 7 day washout period between trials.
Who Masked: Participant, Investigator
Masking Description: Supplements (broccoli seed extract, BSE, and vitamin C (VC) with or without mustard seed powder, MSP) will be in identical capsules, with the double blind code held by the sponsor until after the study is over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broccoli seed extract (Active Comparator): A single dose dietary supplement made up of 385 mg broccoli seed extract delivering 50 mg GR (115 umol GR) and 100 mg vitamin C (as ascorbic acid).
  Interventions: Dietary Supplement: Broccoli seed extract
- Broccoli seed extract with mustard seed powder (Experimental): A single dose dietary supplement made up of a mixture of 385 mg broccoli seed extract delivering 50 mg GR (115 umol GR), 145 mg mustard seed powder containing enough active myrosinase (enzyme) to fully hydrolyze the GR in the capsule to SF post-ingestion (~30 units myrosinase activity) and 100 mg vitamin C (as ascorbic acid).
  Interventions: Dietary Supplement: Broccoli seed extract with mustard seed powder

INTERVENTIONS:
Dietary Supplement: Broccoli seed extract — 2 capsules, one dose
  Arms: Broccoli seed extract
Dietary Supplement: Broccoli seed extract with mustard seed powder — 2 capsules, one dose
  Arms: Broccoli seed extract with mustard seed powder

SUMMARY:
We know that broccoli is a vegetable that is associated with a number of health benefits and is a good choice in a healthy diet. Researchers at major universities, including Johns Hopkins University, have identified nutrients in broccoli that have specific health benefits such as improving antioxidant protection. One of these nutrients is called glucoraphanin (GR). However, in order for GR to deliver health benefits in the human body, it first has to be converted to its active form, sulforaphane (SF). This conversion can happen one of two ways. GR can be converted to SF by our gut bacteria (the microbiota) or it can be converted to SF by an enzyme called myrosinase that is naturally occurring in certain plants, including mustard (the same mustard that is used to make table mustard spread and mayonnaise). The purpose of the present study is to test in healthy human volunteers the oral bioavailability (absorption) of GR in broccoli seed extract (BSE) with or without the presence of active plant myrosinase in mustard seed powder (MSP) delivered in a nutritional supplement.

DETAILED DESCRIPTION:
The aim of the present study is to determine in healthy human volunteers the oral bioavailability of sulforaphane (SF) derived from broccoli seed extract (BSE) standardized to glucoraphanin (GR) content with and without the presence of active plant myrosinase derived from mustard seed powder. Once absorbed, SF is rapidly metabolized by initial conjugation with the endogenous nucleophile glutathione (GSH). The glutathione conjugate then undergoes successive steps of hydrolysis leading ultimately to the formation of the N-acetylcysteine derivatives (mercapturic acids). All of these conjugates are chemically designated dithiocarbamates (DTC) and can be quantified in the blood and urine by mass spectroscopy (MS). Based on previous published studies, it is expected that the conversion of the oral dose of 115 umol of GR to DTC will be about 30-40% (on a molar basis) when GR is co-delivered with mustard seed powder myrosinase, but only 10% when delivered without the myrosinase source. Blood samples will be collected to determine if the supplements influence biomarkers for oxidative stress and inflammation. The stool sample will be used to measure the alpha-diversity of the gut microbiome and whether this has an influence on urine levels of SF and DTC.

This study will include 16 male and female adults ages 25 to 65 years, and employ a randomized crossover design, with a 7 day washout period between trials. Supplements (broccoli seed extract, BSE, and vitamin C (VC) with or without mustard seed powder, MSP) will be in identical capsules, with the double blind code held by the sponsor until after the study is over.

Participants will be recruited and then contacted prior to visit #1 to determine if they match the criteria for entry into the study. Participants will record food and beverages consumed during the evening meal prior to visit #1. Participants will also be instructed to refrain from consuming cruciferous vegetables and condiments that might contain glucosinolates or isothiocyanates (e.g., mustard, horseradish, wasabi, mayonnaise) for 3 days before and during the duration of the study.

Visit #1: Screening, Orientation, Supplementation and Basic Study Procedures Participants will come to the Human Performance Lab (600 Laureate Way, North Carolina Research Campus, Kannapolis, NC) at 7:00, 8:00, or 9:00 am after an overnight fast (at least 9 hours) having avoided consumption of cruciferous vegetables and condiments for at least three days. This visit will begin with a review of the consent form. Height, body weight, body composition (i.e., percent body fat measured on a special scale that participants stand on with bare feet), and blood pressure (automated unit, Omron Healthcare, Inc. Lake Forest, IL, IntelliSense Blood Pressure Monitor Model: HEM-907XL) will be measured in a private section of the lab. The food record for the prior evening meal will be turned in and reviewed with instructions to consume the same meal the evening before Visit #3. Participants will next provide a spot urine sample in a private stall in the restroom. A mid-stream urine sample will be collected in a cup. Next, participants will be randomized to consume 2 capsules containing either BSE + VC or BSE+VC+MSP along with 8 oz. of water. Participants will consume all of the water along with the 2 capsules. The two supplements will be in identical looking capsules so that participants will not be able to determine their identity. Participants and the research will not know which capsules were received at visits 1 or 3 until the study is over. Following intake of the supplement, participants will consume a muffin and coffee within 15 minutes of taking the supplement. Participants will abstain from eating any food or beverages except for water for 2 hours following consumption of the supplement. After the 2-h delay, participants can resume their normal dietary patterns. Participants will collect all urine for the 24 h period after consuming the supplements. Participants will collect all urine for the first 8 hours in one container, and then collect the remaining 8-24 h of urine in a second container. This first visit will take about 1 hour.

Visit #2: Return urine samples and provide blood sample Participants will come to the lab in an overnight fasted state the next morning, drop off the urine collection containers, and provide a blood sample. A stool collection kit with instructions will be given to each participant. (Instructions are included in the forms file attached to this application).

One Day Prior to Visit #3 Participants will collect a small swab sample of stool in a container provided by the lab on Visit #1. Participants will consume the same dinner that was consumed prior to Visit #1.

Visit #3: Supplementation and Basic Study Procedures One week after visit #1, participants will return to the Human Performance Lab at the same time in an overnight fasted state. All the procedures from Visit #1 will be repeated except that participants will consume the opposite supplement.

Visit #4: Return urine samples and provide blood sample Participants (overnight fasted state) will drop off the final urine collection containers at the lab the next morning and provide the fourth and final blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects will be included
* Age between 25-65 years inclusive
* Non-smoker
* Healthy subjects who, in the opinion of the investigator, are free of any medical conditions that might affect study measures
* Body Mass Index (BMI) of 20 - 29.9 kg/m2
* Willingness to adhere to dietary restrictions: refrain from consuming cruciferous vegetables and condiments that might contain glucosinolates or isothiocyanates (e.g., prepared mustard aka deli mustard, mustard greens, horseradish, wasabi, mayonnaise) for 3 days before and for the duration of the study
* Subjects willing to consume the light breakfast consisting of a muffin and 12 oz coffee
* Subjects willing to collect all urine for 24 hours on two separate occasions
* Subjects that have given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Diarrhea or oral antibiotic intake within the last 4 weeks
* Use of proton pump inhibitors (PPIs), antacids or other medications that influence stomach acidity
* Use of laxative medications or other products that promote colon cleansing in the last 4 weeks
* History of malabsorption or GI tract disorders or GI surgeries (i.e. lapband, gastric bypass, etc.)
* Supplementation with broccoli sprout, seed or powder extracts, or other over the counter supplements including the other bioactive ingredients in the test supplement, antioxidants and multi-vitamin mineral supplements, including vitamin C (ascorbic acid), for the previous 2 weeks
* Subject has a known allergy or intolerance to any of the ingredients contained in the test supplements (e.g. broccoli, broccoli seeds, mustard seeds, vitamin C (ascorbic acid))
* Subject is currently pregnant, planning to become pregnant, or is breastfeeding
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Urine concentration of sulforaphane | Change from pre-ingestion to 8- and 24-hours post-ingestion
  Broccoli glucosinolate metabolite

SECONDARY OUTCOMES:
Urine concentration of dithiocarbamate | Change from pre-ingestion to 8- and 24-hours post-ingestion
  Broccoli glucosinolate metabolite

CONTACTS AND LOCATIONS:
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Upon request, will share de-identified data.